CLINICAL TRIAL: NCT04279743
Title: Fatty Acid Metabolism in Carriers of Apolipoprotein E Epsilon 4 Allele: Determining the Blood-to-brain Link
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, Principal investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRSC-2020
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Healthy
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Double-blind controlled randomized study with a parallel study design (40 men and 40 women, ApoE4 carriers and non carriers)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the research nurse will know the randomization of the different treatments administered. All plasma samples collected during the research project will be anonymized i.e. it will not be possible to identify the participant by his name since a number will be assigned to him. The code key linking the participant's name to his number will be stored, with access restricted to those designated by the principal investigator. The data file is also protected by a password.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ApoE4 carriers (Experimental): The results obtained for APOE4 carriers will be compared to the one obtained from APOE4 non-carriers. Carriers are defined as being at least carrier of one APOE4 allele.
  Interventions: Dietary Supplement: omega-3 phospholipids; Dietary Supplement: omega-3 Triglycerides
- ApoE4 non carriers (Experimental): The results obtained for APOE4 carriers will be compared to the one obtained from APOE4 non-carriers. Carriers are defined as being at least carrier of one APOE4 allele.
  Interventions: Dietary Supplement: omega-3 phospholipids; Dietary Supplement: omega-3 Triglycerides

INTERVENTIONS:
Dietary Supplement: omega-3 phospholipids — The intervention is a randomized double blind parallel design testing the metabolism of a krill oil omega-3 phospholipid supplement compared to fish oil omega-3 triglycerides in carriers and non-carriers of the ApoE4 allele. Half of the carriers and non-carriers will receive phospholipids and the other half will receive triglycerides. The intervention choice will be randomized and double blind.
  Participants will be instructed to take 4 supplements every day (2 in the morning and 2 in the evening) (4 g/ day of phospholipids), providing 1.8 g/day of omega-3 fatty acids. They will come back fasted to the research center on weeks 0, 1, 2, 3, 4, 8 and 12 of the study for blood draws. The omega-3 fatty acids metabolism will be compared between the carriers and non carriers of the ApoE4 allele.
Dietary Supplement: omega-3 Triglycerides — The intervention is a randomized double blind parallel design testing the metabolism of a krill oil omega-3 phospholipid supplement compared to fish oil omega-3 triglycerides in carriers and non-carriers of the ApoE4 allele. Half of the carriers and non-carriers will receive phospholipids and the other half will receive triglycerides. The intervention choice will be randomized and double blind.
  Participants will be instructed to take 4 supplements every day (2 in the morning and 2 in the evening), providing 1.8 g/day of omega-3 fatty acids. They will come back fasted to the research center on weeks 0, 1, 2, 3, 4, 8 and 12 of the study for blood draws. The omega-3 fatty acids metabolism will be compared between the carriers and non carriers of the ApoE4 allele.

SUMMARY:
In Canada, ~17 millions of adults between 30-64 y old could benefit from a prevention strategy to lower the risk of Alzheimer's disease (AD). Although a lot of epidemiological studies reported positive cognitive outcomes in populations eating fish, there is skepticism about the link between docosahexaenoic acid (DHA), an omega-3 (OM3) fatty acid in fish and prevention of cognitive decline. This is largely because there is a disconnect between epidemiological, molecular and animal studies which generally favor a link between higher DHA intake and cognition whereas clinical DHA and fish oil trial seem not to support such as link. There are several knowledge gaps in this field that might explain why clinical trials were not successful. This project will focus on two major gaps : OM3 fatty acid metabolism and the blood-to-brain DHA link. OM3 supplements in cardiovascular disease have faced the same issues for decades but the more recent trials have now generated the clinical evidence supporting primary and secondary cardiovascular events reduction and a better risk to benefit balance of OM3 drugs compared to statins, for instance. What if, for cognitive decline, the target was missed because the supplement/drug formulations were not appropriately designed to target the brain? The investigators hypothesize that (i) E4 carriers display a faulty packaging of circulating OM3, leading to reduced bioavailability for brain cells, (ii) The use of new OM3 formulation can direct plasma DHA into brain compartments more readily available for the brain, thereby increasing brain DHA concentrations and improving cognition. Studies in mice and humans will be performed to test OM3 metabolism and the blood-to-brain DHA link. Ultimately the information generated in this research project will help to better design clinical trials in term of fatty acid formulation, expected level to reach in the plasma and the brain.

ELIGIBILITY:
Inclusion Criteria:

- Men and women aged between 30-50 years old.

Exclusion Criteria:

* Tobacco use,
* Malnutrition (assessed from blood albumin, hemoglobin and lipids),
* Diabetes,
* Participants taking an EPA+DHA supplement or consuming more than 2 fish meals per week,
* Uncontrolled thyroid, renal and endocrine disorder disease,
* Chronic immune condition or inflammation (CRP > 10 mg/l, white cell count),
* Cancer,
* Recent major surgery or cardiac event,
* Pregnant or lactating women,
* Pre-menopause or menopause,
* Dementia,
* Ongoing or past severe drug or alcohol abuse,
* Psychiatric difficulties or major depression
* Ongoing or past intensive physical training.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
DHA levels in LPC and FFA | baseline, 1, 2, 3, 4, 8 and 12 weeks after baseline
  To evaluate plasma DHA levels in lysophosphatidylcholine and free fatty acids by ApoE genotype and treatment intervention.
EPA levels in LPC and FFA | baseline, 1, 2, 3, 4, 8 and 12 weeks after baseline
  To evaluate plasma EPA levels in lysophosphatidylcholine and free fatty acids by ApoE genotype and treatment intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Plourde, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No